CLINICAL TRIAL: NCT05633082
Title: A Clinical Performance of Two Soft Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-143
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-11

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: All participants received Lens 1 and then Lens 2 in fixed-sequence order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens 1 (Experimental): All participants wore Lens 1 for 15 minutes (Period 1)
  Interventions: Device: Lens 1 (omafilcon B)
- Lens 2 (Experimental): All participants wore Lens 2 for 15 minutes (Period 2)
  Interventions: Device: Lens 2 (fanfilcon A)

INTERVENTIONS:
Device: Lens 1 (omafilcon B) — Toric daily wear contact lens for 15 minutes
  Arms: Lens 1
Device: Lens 2 (fanfilcon A) — Toric daily wear contact lens for 15 minutes
  Arms: Lens 2

SUMMARY:
The study objective was to gather short-term clinical performance data for two soft toric contact lenses.

DETAILED DESCRIPTION:
This participant-masked, non-randomized, controlled non-dispensing study was to compare the performance of two soft toric lenses. Participants attended one study visit which lasted for approximately 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* They are of legal age (18) and capacity to volunteer.
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They currently wear soft contact lenses, or have done so within the past two years.
* They have ocular astigmatism in both eyes of between 0.75DC and 3.00DC.
* They are expected to be able to be fitted with the study lenses within the power range available.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They are aphakic.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or lactating.
* They have an eye or health condition including an immunosuppressive or infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or a history of anaphylaxis or severe allergic reaction.
* They have taken part in any contact lens or care system clinical research within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD, MCOptom, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens 1 (Omafilcon B): All participants wore Lens 1 for 15 minutes (Period 1)
- Lens 2 (Fanfilcon A): All participants wore Lens 2 for 15 minutes (Period 2)
Period: Period 1: Lens 1, 15 Minutes
Arm/Group | Lens 1 (Omafilcon B) | Lens 2 (Fanfilcon A)
Started | 40 | 0 (All participants received Lens 1 in Period 1.)
Completed | 40 | 0
Not Completed | 0 | 0
Period: Period 2: Lens 2, 15 Minutes
Arm/Group | Lens 1 (Omafilcon B) | Lens 2 (Fanfilcon A)
Started | 0 (All participants received Lens 2 in Period 2.) | 40
Completed | 0 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes all study participants.
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Score
Description: The subjective overall impression of the contact lens (scored as a single value per participant) was assessed using a 0-100 visual analogue scale where 0=Extremely poor, 100=Excellent.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens 1: Participants that received Lens 1
- Lens 2: Participants that received Lens 2
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 40 | 40
score on a scale | 71.6 (20.2) | 78.9 (16.2)

2. Secondary Outcome: Subjective Comfort
Description: Subjective comfort (scored as a single value per participant) was assessed using a 0-100 visual analogue scale where 0=Causes pain,100=Excellent.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 40 | 40
score on a scale | 74.6 (19.5) | 85.0 (15.0)

3. Secondary Outcome: Subjective Vision
Description: Subjective vision (scored as a single value per participant) was assessed using a 0-100 visual analogue scale where 0=Unacceptable,100=Excellent.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 40 | 40
score on a scale | 76.6 (19.4) | 78.8 (16.6)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 1.5 hours.
Arm/Group | Lens 1 | Lens 2
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05633082/Prot_SAP_000.pdf